CLINICAL TRIAL: NCT04588545
Title: Phase I/II Study of Radiation Therapy Followed by Intrathecal Trastuzumab/Pertuzumab in the Management of HER2+ Breast Leptomeningeal Disease
Brief Title: Radiation Therapy Followed by Intrathecal Trastuzumab/Pertuzumab in HER2+ Breast Leptomeningeal Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20487; ML41590 (Other: Genetech)
Record Dates: First submitted 2020-10-07; First posted 2020-10-19 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: HER2-positive Breast Cancer; Leptomeningeal Metastasis; Leptomeningeal Disease
MeSH Terms: conditions — Meningeal Carcinomatosis; Meningeal Neoplasms | interventions — Radiotherapy; pertuzumab; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Radiation Therapy followed by 10 mg Pertuzumab and 80 mg Trastuzumab (Experimental): Treatment will be initiated with radiation therapy (RT), either whole brain radiation therapy or focal brain/spine radiation therapy. Participants will be treated at dose level 1 of 4 with 10 mg pertuzumab along with 80 mg trastuzumab via Ommaya reservoir over 2-5 minutes. Pertuzumab and trastuzumab will be administered sequentially. Participants will be observed 30 to 60 minutes before commencing the next agent. Participants will be treated twice a week for 4 weeks, once a week for 4 weeks, and then once every 2 weeks.
  Interventions: Radiation: Radiation Therapy; Drug: Pertuzumab; Drug: Trastuzumab
- Radiation Therapy followed by 20 mg Pertuzumab and 80 mg Trastuzumab (Experimental): Treatment will be initiated with radiation therapy (RT), either whole brain radiation therapy or focal brain/spine radiation therapy. Participants will be treated at dose level 2 of 4 with 20 mg pertuzumab along with 80 mg trastuzumab via Ommaya reservoir over 2-5 minutes. Pertuzumab and trastuzumab will be administered sequentially. Participants will be observed 30 to 60 minutes before commencing the next agent. Participants will be treated twice a week for 4 weeks, once a week for 4 weeks, and then once every 2 weeks.
  Interventions: Radiation: Radiation Therapy; Drug: Pertuzumab; Drug: Trastuzumab
- Radiation Therapy followed by 40 mg Pertuzumab and 80 mg Trastuzumab (Experimental): Treatment will be initiated with radiation therapy (RT), either whole brain radiation therapy or focal brain/spine radiation therapy. Participants will be treated at dose level 3 of 4 with 40 mg pertuzumab along with 80 mg trastuzumab via Ommaya reservoir over 2-5 minutes. Pertuzumab and trastuzumab will be administered sequentially. Participants will be observed 30 to 60 minutes before commencing the next agent. Participants will be treated twice a week for 4 weeks, once a week for 4 weeks, and then once every 2 weeks.
  Interventions: Radiation: Radiation Therapy; Drug: Pertuzumab; Drug: Trastuzumab
- Radiation Therapy followed by 80 mg Pertuzumab and 80 mg Trastuzumab (Experimental): Treatment will be initiated with radiation therapy (RT), either whole brain radiation therapy or focal brain/spine radiation therapy. Participants will be treated at dose level 4 of 4 with 80 mg pertuzumab along with 80 mg trastuzumab via Ommaya reservoir over 2-5 minutes. Pertuzumab and trastuzumab will be administered sequentially. Participants will be observed 30 to 60 minutes before commencing the next agent. Participants will be treated twice a week for 4 weeks, once a week for 4 weeks, and then once every 2 weeks.
  Interventions: Radiation: Radiation Therapy; Drug: Pertuzumab; Drug: Trastuzumab

INTERVENTIONS:
Radiation: Radiation Therapy — Participants will receive radiation therapy (RT), either whole brain radiation therapy or focal brain/spine RT. The goal of RT is to palliate symptoms and improve the flow of Intrathecal (IT) therapy through the cerebrospinal fluid (CSF). As such, various RT schedules and targets are permitted. It is expected that the majority of patients will receive WBRT with 30 Gy in 10 fractions. However, shorter fractions of 20 Gy in 5 fractions of WBRT are permitted. In those patients who have more localized leptomeningeal disease in the spine, focal RT in up to 10 fractions may be administered with the exact dose left up to the discretion of the treating radiation oncologist.
Drug: Pertuzumab — Participants will be treated at 1 of 4 dose levels of pertuzumab, beginning at 10 mg and increasing up to 80 mg or Maximum Tolerated Dose (MTD).
Drug: Trastuzumab — Participants will be treated at a fixed dose of 80 mg trastuzumab.

SUMMARY:
The purpose of this study is to find out if radiation therapy followed by intrathecal trastuzumab and pertuzumab is safe and will result in improved survival in HER2 positive breast cancer which has metastasized to the leptomeninges.

DETAILED DESCRIPTION:
The study is designed as a prospective, single-arm, nonrandomized, open-label, phase I/II trial of radiation therapy (RT) followed by intrathecal (IT) trastuzumab/pertuzumab in the management of HER2+ breast leptomeningeal disease (LMD). Treatment will be initiated with RT, whole brain RT (WBRT) and/or focal brain/spine RT followed by IT trastuzumab/pertuzumab.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of HER2 positivity. All patients with HER2+ cancers will be allowed to enroll if they have leptomeningeal disease (LMD). Patients may be IHC 3+ and/or FISH-positive. IHC 2+ HER2 patients are eligible with reflex FISH-positive testing with the ratio ≥2.0.

And/or patients with HER2 positive cells in the cerebral spinal fluid.

* Participants may have concomitant brain metastases
* Cerebrospinal fluid (CSF) sampling is required to document LMD if not documented by MRI. Participants are still eligible CSF is negative but LMD disease is documented on MRI
* Life expectancy greater than 8 weeks
* Consent to pretreatment tumor biopsy or retrieval of archival tissue
* Normal renal (creatinine <1.5 × upper limit of normal [ULN]), liver (bilirubin < 1.5 × ULN, transaminases <3.0 × ULN, except in known hepatic disease, wherein may be <5 × ULN) and blood counts (white blood cells ≥2.5, neutrophils ≥1000, platelets ≥75,000, hemoglobin ≥8)
* LVEF >50%
* KPS >/= 60
* Patients with surgery within 14 days should have recovered from all effects of the surgery and be cleared by their surgeon
* There is no limit on prior systemic or IT therapies
* Must be willing to have an Ommaya reservoir placed and a candidate for an Ommaya reservoir placement
* Women of childbearing potential and sexually active males must commit to the use of effective contraception while on study. Contraception methods should start a minimum of 14 days before the first administration of study drug and continue for the duration of study treatment and for at least 7 months after the last dose of study treatment.
* Ability to sign informed consent.
* Patients may continue treatment with IV trastuzumab, pertuzumab, or other HER2-directed, hormonal, or chemotherapeutic agents if controlling systemic disease and leptomeningeal metastases that developed while on these therapies. In addition, at time of systemic progression, patients may start additional agents at the discretion of the treating physician according to criteria per protocol.

Exclusion Criteria:

* Current or prior participation in a study of an investigational agent or investigational device within 2 weeks of the first dose of study treatment
* Cannot be on systemic agents (chemotherapy) that have Central Nervous System (CNS) penetration (temozolomide, carmustine, lomustine, etoposide, capecitabine, carboplatin, vinorelbine, bevacizumab, irinotecan, and topotecan) unless they develop or have progressive or persistent leptomeningeal metastases while on these agent(s). See protocol for additional information regarding systemic therapies.
* Major surgery or significant traumatic injury that has not been recovered from 14 days before the initiation of study drug
* Symptomatic lung disease resulting in shortness of breath at rest
* Women who are pregnant or breastfeeding
* History of serious adverse event to any of the study drugs or study drug components
* Whole Body Radiation Therapy (WBRT) is not allowed while patients receive IT trastuzumab/pertuzumab; however, focal stereotactic or palliative RT is allowed
* Significant medical or psychiatric illness that would interfere with compliance and ability to tolerate treatment as outlined in the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Maximum Tolerated Dose (MTD) of Intrathecal (IT) pertuzumab in combination with IT trastuzumab | Up to 12 weeks per dosing cohort
  MTD will be determined by testing increasing doses or pertuzumab beginning at 10 mg increasing to 20 mg, 40 mg and 80 mg, along with a fixed dose of 80 mg Trastuzumab.
Phase 2: Overall Survival (OS) | 1 year after study enrollment
  1 year Overall Survival (OS), defined as the time between the date of study enrollment and the date of death due to any cause.

SECONDARY OUTCOMES:
Response Rate | Up to 1 year
  All patients included in the study will be assessed for response to treatment. Each patient will be assigned one of the following categories: 1) Complete Response,2) Partial Response, 3) Stable Disease, 4) Progressive Disease, 5) Early death due to disease, 6) Early death due to toxicity 7)Early death due to unknown cause. Participants in categories 4 through 6 would be considered as failing to respond to treatment.
Progression Free Survival (PFS) | Up to 1 year
  PFS measured from the date of first treatment to the date of first observation of Progressive Disease (PD), nonreversible neurologic progression, or death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Ahmed, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Northwestern University, Evanston, Illinois

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Moffitt Cancer Center's Clinical Trials Website — https://moffitt.org/clinical-trials-research/clinical-trials/